CLINICAL TRIAL: NCT05166785
Title: BRInging the Diabetes Prevention Program to GEriatric Populations
Acronym: BRIDGE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-01039; 1R01DK127916-01A1 (NIH)
Record Dates: First submitted 2021-12-08; First posted 2021-12-22 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Pre Diabetes
MeSH Terms: conditions — Glucose Intolerance | interventions — Aging

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-person Diabetes Prevention Program (DPP) (Active Comparator): Participants randomized to the in-person DPP intervention for 12 months
  Interventions: Other: In-Person Diabetes Prevention Program (DPP)
- DPP program Tailored for Older Adults and delivered via Telehealth (DPP-TOAT arm) (Active Comparator): Participants randomized to the DPP program Tailored for Older Adults and delivered via Telehealth (DPP-TOAT arm) intervention for 12 months.
  Interventions: Other: DPP Tailored for Older Adults and delivered via Telehealth

INTERVENTIONS:
Other: DPP Tailored for Older Adults and delivered via Telehealth — Diabetes Prevention Program (DPP) Tailored for Older Adults and delivered via Telehealth (DPP-TOAT) will be composed of 16 60-minute weekly sessions followed by six 60-minute monthly support sessions
  Arms: DPP program Tailored for Older Adults and delivered via Telehealth (DPP-TOAT arm)
Other: In-Person Diabetes Prevention Program (DPP) — Diabetes Prevention Program (DPP) is composed of 16 60-minute weekly sessions followed by six 60-minute monthly support sessions over 12 months in person approved by the Centers for Disease Control and Prevention (CDC)
  Arms: In-person Diabetes Prevention Program (DPP)

SUMMARY:
Over 24 million Americans are over 65 years and have prediabetes. Prediabetes can be addressed using a public health approach: among the 20% of participants in the Diabetes Prevention Program (DPP) who were ages 60 and over, the diet and physical activity intervention conferred a 71% risk reduction of diabetes after an average follow-up of 3 years. The population of older adults is projected to more than double from 52.5 million in 2019 to ~100 million by 2060, and if projections hold, about half (48.3%) will have prediabetes. The proposed hybrid effectiveness implementation type 1 design will compare a DPP program Tailored for Older Adults and delivered via Telehealth (DPP-TOAT arm) to an in person DPP tailored for older adults (DPP arm) using a randomized, controlled trial design (n=230). The preliminary data suggests DPP-TOAT is a feasible and acceptable way to deliver the DPP to older adults, and this will be the first study to compare the effectiveness and implementation of two strategies (telehealth versus in-person) to deliver a tailored DPP for the unique needs of the growing population of older adults.

DETAILED DESCRIPTION:
Eligible patients will be recruited through electronic health records (Epic and MyChart) and randomized to the 12-month DPP-TOAT or the in-person DPP program. Primary effectiveness outcome will be 6-month weight loss and implementation outcome will be attendance. A pragmatic approach will be used in order to inform future studies conducted in community-based and rural settings. Findings will inform best practices in the delivery of an evidence-based intervention that could reach the 30+ million adults aged 65 and over with prediabetes.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 65 years and older
* Diagnosis of pre-diabetes (A1c between 5.7-6.4%, fasting glucose between 100-125 mg/dL, or oral glucose tolerance test between 140-199 mg/dL within past 12 months)
* BMI of greater than or equal to 30
* English-speaking
* Under the care of a Primary care provider (PCP) in the NYU Langone Health system
* Able to travel to NYU Langone for in-person evaluations
* Access to a telephone
* Informed consent

Exclusion Criteria:

* Prevalent diabetes or end-stage renal disease
* Prior participation in the Diabetes Prevention Program
* A documented current history of active psychosis or other cognitive issues via International Classification of Diseases (ICD) -10 codes
* Taking FDA-approved weight loss medications
* PCP stating that patient should not participate
* Inability to communicate due to severe, uncorrectable hearing loss or speech disorder
* Severe visual impairment that precludes completion of assessments and/or intervention

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 238 (Actual)
Dates: Start 2022-10-05 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Changes in weight in participants in DPP-TOAT is similar to those in In-Person DPP | Baseline visit, 6 months visit, 12 month visit
  In-person outcome assessment visits at the New York University Langone research clinic to measure weight at baseline, 6, and 12 months among all randomized participants
Changes in HbA1c in participants in DPP-TOAT is similar to those in In-Person DPP | Baseline visit, 6 months visit, 12 month visit
  In-person outcome assessment visits at New York University Langone research clinic to measure glycemia at baseline, 6, and 12 months among all randomized participants

SECONDARY OUTCOMES:
Adherence to the DPP-TOAT is greater than the in-person DPP | Baseline visit, 6 months visit, 12 month visit
  This will be measured by the number of group sessions completed by each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Jeannette M Beasley, PhD, RDN, Principal Investigator — NYU Langone Health; Joshua Chodosh, MD, MHS, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Data collected from this study include anthropometric and blood draw data that will be uploaded to the participants' electronic medical record and questionnaire data that will only be used for study-related purposes.

DOCUMENTS (1):
  • Informed Consent Form (2022-12-02): https://cdn.clinicaltrials.gov/large-docs/85/NCT05166785/ICF_000.pdf